CLINICAL TRIAL: NCT05772806
Title: Diagnostic Approach of Early Atrial Fibrillation, Silent Stroke and Cognitive Disorder in Patients With High-risk: Multicenter, Prospective Cohort Study
Brief Title: Diagnostic Approach of Early Atrial Fibrillation, Silent Stroke and Cognitive Disorder in Patients With High-risk
Acronym: PREFA-TE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Català de la Salut (Other)
Responsible Party: Sponsor
Other Study IDs: SLT/21/000027
Record Dates: First submitted 2023-02-22; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2022-12

CONDITIONS: Atrial Fibrillation; Atrial Fibrillation New Onset; Dementia; Stroke
Keywords: Atrial Fibrillation; Dementia; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Dementia; Stroke | interventions — Electrocardiography; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood plasma and serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Electrocardiogram — The electrocardiogram will help to diagnose atrial fibrillation and the electronic devices (App Fibricheck and Smart bracelet/watch) will help to detect an arrhythmic rhythm.
  The echocardiography will be used for detecting criteria of atrial cardiomyopathy.
  MRI may help to detect silent strokes.
  Other Names: echocardiography, MRI, Smart Bracelet/watch, Fibricheck

SUMMARY:
The goal of this observational study is to determine the impact of the combined use of cardiac rhythm recording devices, biomarkers, echocardiogram, and Magnetic Resonance Imaging (MRI) on the early detection of AF, silent stroke, and cognitive impairment in subjects older than 65 years at high risk.

The main questions it aims to answer are:

* The early detection of AF, allowing the establishment of preventive measures, will avoid its main complications, especially strokes and cognitive impairment or dementia, in patients at high risk?
* Will cardiac rhythm monitoring devices be useful in the early detection of AF in patients at high risk? Participants will undertake an initial evaluation through an echocardiogram (to detect atrial dysfunction), cranial MRI (to detect silent strokes), plasma/serum collection to determine biomarkers, and a complete clinical assessment (including electrocardiogram, and scales for measurement of cognitive and functional status). The clinical evaluation will be repeated every 6 months and will allow the recording of the date of occurrence of the study events. In addition, annually, patients will be subjected to cardiac rhythm monitoring by electronic devices with the aim of improving AF detection.

DETAILED DESCRIPTION:
Design: Multicenter, prospective cohort study Setting and study population: Patients will be recruited from the usual consultations in six Primary Health Care Centers (PHCC) managed by the Catalan Health Institute (ICS), two in Tarragonés county and four in Terres de l'Ebre county, both situated in Tarragona (South Catalonia, Spain).

Study subjects: Patients between 65-85 years old at high risk of FA who are attended at study' PHCCs, consent to participate, and meet inclusion criteria.

Follow-up: Initially all included patients will undertake echocardiography, biomarkers, and cranial /brain Magnetic resonance imaging (MRI). Cardiac monitoring (for 14 days) with two different electronic devices will be performed once every year during the study period. Every six-month electrocardiogram and complete clinical assessment will be done to register risk factors and comorbidities, new cardiovascular events, anthropometric parameters (arterial pressure, heart rate…), and scores at different tests related to functional status (Barthel or Rankin), cognitive function (Global Deterioration Scale [GBS], Mini-Mental State Examination [MMSE]), or AF / stroke risk (CHADsVASc, HAS-BLED). Any changes in the electronic prescription made by the professional according to the patient's assessment will also be recorded.

Data recording: Most of the study data will be recorded from evaluations/tests performed on patients (from anamnesis -including scales-, physical examination, and laboratory tests) or reports provided by specialists (available at computerized clinical history [e-SAP]), in the case of echocardiography (cardiologist) or MRI (radiologist) searching especially atrial dysfunction and signs of silent strokes. Data registered in the electronic primary care health records (e-CAP) of participants will also be collected. Therapeutic (pharmacological) changes will be registered from the SIRE (Catalan acronym for Integrated Electronic Prescription System). Finally, cardiac monitoring data will be collected through the electronic devices' registers. An ad hoc data collection questionnaire will be created to register and store all study variables. The electronic questionnaire will be available at a specific application (where data will remain stored for five years) accessible from the corporate (ICS) Intranet; only study researchers, through personal passwords, may record and access data.

Definition of the outcome variable: Time until the diagnosis of atrial fibrillation (confirmed by electrocardiogram), stroke (new diagnosis in e-CAP or confirmed by neuroimaging) , and cognitive impairment/dementia [diagnosed through Score in Global Deterioration Scale (GDS)].

Sample calculation: To detect a difference of 0.1 units in the prevalence of atrial fibrillation observed, compared to the reference (0.07) accepting an alpha risk of 0.05 and a beta risk of 0.05 a sample of 148 individuals will be required. Estimated loss rate at 15 per cent.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 65-85 years old
* Patients in Q4 (highest risk) of Atrial Fibrillation (AF). [Clua-Espuny et al, 2020]
* CHADsVASc ≥ 2
* Being capable of using a Smart phone (or the care giver)

Exclusion Criteria:

* Patients with previous diagnostic of AF, stroke, or dementia.
* Patients treated with anticoagulants.
* Vital prognosis less than one year.
* Severe cognitive or functional impairment (GDS ≥ 3, and/or Barthel score ≤60, or MRS Rankin ≥4, or severe mobility impairment)
* Pacemaker Carrier

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients between 65-85 years old at high risk of AF will be recruited from the usual consultations in six Primary Health Care Centers (PHCC) managed by the Catalan Health Institute (ICS), two in Tarragonés county and four in Terres de l'Ebre county , both situated in Tarragona (South Catalonia, Spain).
Sampling Method: Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Atrial Fibrillation | Through study completion, an average of 2 years
  New diagnoses of atrial fibrillation could be made during protocolized evaluations every six months (including electrocardiography) or at any time during the study period, provided that an electrocardiogram is performed on the participant, on suspicion of arrhythmia or for any other reason.
  Moreover, a search for new-onset atrial fibrillation will be undertaken for 14 days twice during the study period, through cardiac monitoring with smart bracelets (constant monitoring) and using the FibriCheck application (two times a day and in case of symptoms). All new AF diagnoses will require confirmation via 12-lead electrocardiogram
Stroke | Through study completion, an average of 2 years
  Silent strokes may be detected through cranial MRI at initial evaluation. During the study period new stroke diagnoses will require confirmation through a neuroimaging test or neurologist assessment.
Cognitive impairment/ Dementia | Through study completion, an average of 2 years
  Cognitive impairment will be assessed through changes in the Global Deterioration Scale (GDS) score; scores from four will be considered diagnoses of dementia. This diagnosis will also be considered if confirmed through the neurologist's evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Lluís Clua-Espuny, MD PhD, Principal Investigator — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina; Eva Maria Satue-Gracia, MD PhD, Study Director — Institut Català de la Salut; Francisco M. Martín-Luján, MD PhD, Study Director — University Rovira i Virgili
Locations (1):
- Eva Maria Satue Gracia, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: Yes
not yet decided as future studies are being considered and may be considered
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 years
Access Criteria: The data will be entered on the IDIAP J Gol institution platform
URL: http://www.idiapjgol.org/index.php/ca/

REFERENCES:
- [Derived] Hernandez-Pinilla A, Clua-Espuny JL, Satue-Gracia EM, Palleja-Millan M, Martin-Lujan FM; PREFA-TE Study-Group. Protocol for a multicentre and prospective follow-up cohort study of early detection of atrial fibrillation, silent stroke and cognitive impairment in high-risk primary care patients: the PREFA-TE study. BMJ Open. 2024 Feb 19;14(2):e080736. doi: 10.1136/bmjopen-2023-080736. PMID 38373864